CLINICAL TRIAL: NCT00206219
Title: A Phase III Randomised, Stratified, Parallel-Group, Multi-Centre, Comparative Study of ZD1839 (Iressa®) 250 Mg and 500 Mg Versus Methotrexate for Previously Treated Patients With Squamous Cell Carcinoma of the Head and Neck
Brief Title: Head and Neck Phase III Iressa Versus Methotrexate Refractory: Iressa Versus Methotrexate (IMEX)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0704; EudraCT no.2004-002662-38; NCT00072878 (obsolete NCT alias)
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Gefitinib; Methotrexate

INTERVENTIONS:
Drug: Gefitinib
Drug: methotrexate

SUMMARY:
This study is to compare ZD1839 (250mg and 500mg) versus methotrexate in head and neck cancer in terms of overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of evidence of squamous cell carcinoma of the head and neck.
* Tumors have progressed after primary treatment with radiation or chemoradiation and have failed to respond to at least one course of standard platinum-based chemotherapy.
* Tumors have progressed after primary treatment with radiation or chemoradiation and are considered unsuitable for platinum-based chemotherapy.

Exclusion Criteria:

* Carcinomas of the post-nasal space, thyroid, sinus or salivary gland tumors.
* Isolated recurrent disease that may be amenable to local therapy; e.g., surgical intervention or radiation therapy.
* Known severe hypersensitivity to ZD1839, Methotrexate or any of the excipients of these products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477
Dates: Start 2003-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Compare ZD1839 versus methotrexate in overall survival

SECONDARY OUTCOMES:
Compare ZD1839 versus methotrexate in symptom improvement, tumor response, safety and tolerability and quality of life - assessed throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (109):
- United States (26):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Palm Springs, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Norwalk, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormand Beach, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Des Moines, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Waterville, Maine
  - Research Site, Bethesda, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Hackensack, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Norfolk, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (4):
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, El Palomar, Buenos Aires
  - Research Site, Salta, Salta Province
  - Research Site, Santa Fe, Santa Fe Province
- Research Site, Westmead, New South Wales, Australia
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Haine-Saint-Paul
- Brazil (3):
  - Research Site, Goiânia, Goiás
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, São Paulo, São Paulo
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Zagreb, Croatia
- Czechia (4):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Ostrava - Poruba
  - Research Site, Prague
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Research Site, Thessaloniki, Greece
- India (8):
  - Research Site, Kochi, Kerala
  - Research Site, Thiruvananthapuram, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Pune, Maharashtra
  - Research Site, Ansārinagar, New Dehli
  - Research Site, Jaipur, Rajasthan
  - Research Site, Kolkata, West Bengal
  - Research Site, New Dehli
- Israel (2):
  - Research Site, Petah Tikva
  - Research Site, Tel Litwinsky
- Italy (8):
  - Research Site, Bologna
  - Research Site, Cuneo
  - Research Site, Forlì
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Torino
- Research Site, Riga, Latvia
- Lithuania (2):
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Malaysia (2):
  - Research Site, Kampung Baharu Nilai
  - Research Site, Petaling Jaya
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Utrecht
- Research Site, Oslo, Norway
- Russia (3):
  - Research Site, Krasnogorsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovenia (2):
  - Research Site, Zaloska, Ljubljana
  - Research Site, Ljubljana
- South Africa (6):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pretoria
  - Research Site, Tygerberg
- Spain (10):
  - Research Site, Santiago de Compostela, A Coruña
  - Research Site, Granada, Granada
  - Research Site, Leganés, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Pontevedra, Pontevedra
  - Research Site, Valencia, Valencia
  - Research Site, Barakaldo, Vizcaya
  - Research Site, Santander
  - Research Site, Valencia
  - Research Site, Vitoria-Gasteiz, Álava
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
- United Kingdom (2):
  - Research Site, Leeds
  - Research Site, London